CLINICAL TRIAL: NCT03986671
Title: A Pilot Study to Assess Transmembrane Electromyography (TM-EMG) for the Assessment of Neuromuscular Function in the Oropharynx
Brief Title: Transmembrane Electromyography (TM-EMG) for the Assessment of Neuromuscular Function in the Oropharynx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Powell Mansfield Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TM-EMG Pilot Study
Record Dates: First submitted 2019-05-22; First posted 2019-06-14 (Actual); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Obstructive Sleep Apnea; Amyotrophic Lateral Sclerosis; Muscular Dystrophies; Healthy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Amyotrophic Lateral Sclerosis; Muscular Dystrophies

STUDY DESIGN:
Intervention Model Description: This is a prospective, cohort, pilot study with blinded data analysis and two physician testers to assess intertester reliability and device usability. Volunteers will include healthy adults, participants with documented neurologic pharyngeal muscle dysfunction (ALS and muscular dystrophy), and participants with severe OSA. For each participant diagnostic properties of EMG studies will be assessed using a conventional needle and TM-EMG sensor in pharyngeal muscles.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- EMG Testing (Experimental): Examination of the electromyographic signal from oropharyngeal muscles obtained using an investigational transmenbrane sensor attached to a rigid probe and an FDA-approved very fine concentric needle electrode (Ambu Neuroline 25 mm x 30G).
  Interventions: Device: Transmembrane EMG Oropharynx Probe

INTERVENTIONS:
Device: Transmembrane EMG Oropharynx Probe — Examination of the electromyographic signal from oropharyngeal muscles obtained using an investigational transmembrane sensor attached to a rigid probe and an FDA-approved very fine concentric needle electrode (Ambu Neuroline 25 mm x 30G).

SUMMARY:
This is a pilot study to examine the diagnostic utility of a novel transmembrane surface sensor, and compare signals obtained with the transmembrane sensor to conventional needle EMG signals from healthy volunteers to those with documented neurologic pharyngeal muscle dysfunction (ALS and muscular dystrophy) and to those with severe OSA.

DETAILED DESCRIPTION:
Transmembrane electromyography (TM-EMG) may be a feasible and valid non-invasive EMG technique for detecting neuromuscular (NM) impairment. This study will assess whether, in healthy volunteers and participants with known obstructive sleep apnea (OSA) and other NM diseases involving the oropharynx, the same characteristic motor unit potentials obtained on conventional needle EMG (NEMG) can be obtained using a TM-EMG sensor. The purpose of this study is to demonstrate whether the TM-EMG sensor can provide the same diagnostic accuracy as the concentric needle electrode for the diagnosis of NM diseases. Having demonstrated diagnostic similarity of TM-EMG to NEMG, the secondary aim of this study is to confirm that NM disturbance of oropharyngeal striated muscles in participants with OSA can be elicited with the TM-EMG sensor.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* Must be able to pause use of anticoagulation, NSAID and multi-vitamins for appropriate period prior to study test.
* Must be willing to stop any type of smoking or vaping 10 days prior to testing

A cohort of participants with documented neurological disorders involving upper airway striated muscles including ALS and muscular dystrophy with the presence of bulbar symptoms.

A cohort of participants diagnosed with moderate to severe OSA proven by an in-lab PSG, including the following criteria:

* AHI > 25
* Nadir SaO2 < 85%
* not currently using CPAP

A cohort of healthy participants that meet the following criteria:

* Normal craniofacial anatomy
* BMI < 30

Exclusion Criteria:

* Allergy to topical anesthetic
* 4 or more alcoholic drinks on the same occasion on 5 or more days in the past month
* Prior cancer, or radiation to the head or neck
* Craniofacial anatomical disorders
* Presence of any underlying medical, surgical or psychiatric disorder that would preclude participation as determined by the principal investigator

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-04-30 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Perry Mansfield, MD, Principal Investigator — Perry Mansfield MD Inc.
Locations (1):
- SENTA Clinic, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Normal Subjects: A group of subjects that have been confirmed to have normal oropharyngeal anatomy by an ENT, and also had an overnight in lab PSG with an AHI < 2.
- Amyotrophic Lateral Sclerosis: Patients having a confirmed diagnosis of Amyotrophic Lateral Sclerosis (ALS) with bulbar involvement.
- Obstructive Sleep Apnea (OSA): Subjects with a confirmed diagnosis of OSA confirmed by in-laboratory polysomnography (PSG) with an AHI of 25 or higher.
Period: Overall Study
Arm/Group | Normal Subjects | Amyotrophic Lateral Sclerosis | Obstructive Sleep Apnea (OSA)
Started | 36 | 9 | 5
Passed a Screening Visit With ENT | 6 | 5 | 5
Completed | 6 | 5 | 5
Not Completed | 30 | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Normal Subjects | Amyotrophic Lateral Sclerosis | Obstructive Sleep Apnea (OSA) | Total
Number analyzed (Participants) | 6 | 5 | 5 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 3 | 12
  >=65 years | 0 | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.66 (3.90) | 59.20 (11.63) | 53.20 (11.41) | 45.47 (18.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 1 | 8
  Male | 1 | 3 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Proof of Diagnostic Consistency
Description: Proof of diagnostic consistency using both the TM-EMG sensor and NEMG in neuromuscular disorders of the oropharyngeal muscles. Significant Inter rater reliability between two blinded neuromuscular experts when using TM-EMG in the palatoglossal and genioglossus.
Time Frame: 1 hour
Measure: Number; unit: % agreement
Groups:
- Obstructive Sleep Apnea (OSA): Subjects with a confirmed diagnosis of moderate to severe OSA confirmed by in-laboratory polysomnography (PSG) with an AHI of 25 or higher.
Arm/Group | Normal Subjects | Amyotrophic Lateral Sclerosis | Obstructive Sleep Apnea (OSA)
Number analyzed (Participants) | 6 | 5 | 5
% agreement | 95.7 | 78.1 | 90

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: Same Definition as clinicaltrials.gov
Arm/Group | Normal Subjects | Amyotrophic Lateral Sclerosis | Obstructive Sleep Apnea (OSA)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03986671/Prot_SAP_000.pdf